CLINICAL TRIAL: NCT05237700
Title: Symptoms, Functional Status and Quality of Life in Patients Undergoing Robotic-assisted and Laparoscopic Surgery in Steep Trendelenburg With or Without Lithotomy Positioning on the Operating Table.
Brief Title: Steep Trendelenburg With or Without Lithotomy Positioning on the Operating Table.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Signe Berit Bentsen, Professor, registered nurse, operating room nurse, Oslo University Hospital
Other Study IDs: 104764
Record Dates: First submitted 2022-01-20; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Neuropathy; Intraoperative Injury; Intraoperative Complications; Patient Positioning; Operating Table
MeSH Terms: conditions — Peripheral Nervous System Diseases; Intraoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trendelenburg with lithotomy positioning on the operating table.: The patient is positioned in Trendelenburg with lithotomy positioning on the operating table.
  Interventions: Other: Patient positioning on operating table
- Trendelenburg without lithotomy positioning on the operating table.: The patient is positioned in Trendelenburg without lithotomy positioning on the operating table.
  Interventions: Other: Patient positioning on operating table

INTERVENTIONS:
Other: Patient positioning on operating table — The patients are either positioned in Trendelenburg with lithotomy positioning or in Trendelenburg without lithotomy positioning on the operating table when undergoing robotic assisted laparoscopic surgery or laparoscopic surgery.

SUMMARY:
Robotic assisted laparoscopic and laparoscopic gynecological, colon-rectal and urological surgical procedures require that patients be placed in steep Trendelenburg positioning with or without lithotomy on operating table. Steep Trendelenburg positioning is a variation of supine positioning in which the patient lies face up with the head and body tilted 250-450 downwards. In lithotomy position the legs are placed in stirrups and knees bent flexing the leg on the operating table. Lithotomy position can be graded in four levels according to what access the surgeon needs. The arms are tucked and padded parallel to the body, or the arms left on an arm board at an angel of less 900. Intraoperative peripheral nerve injury (IPNI) may follow incorrect positioning, inadequate fixation, or prolonged time in positioning. IPNI is defined as new (within 48 h) sensory and/or motor deficits and occurs following a combination of stretch, ischemia and/or compression during surgery and the injuries are either temporary or permanent. In a systematic review we found that IPNI was related to lithotomy positioning with steep Trendelenburg in upper and lower extremity and the incidence of IPNI ranges from 0.16% to 10 %. IPNI after patient positioning on operating table has been described to result in pain and other symptoms as numbness, weakness, and tingling. As demonstrated in our systematic review many of the patients with IPNI did not report pain, which also supported in a recent review. In addition, our systematic review showed that the symptoms appeared immediately after surgical procedures and usually subside within three months. The systematic review also demonstrates that a few patients continue to have pain or/and other symptoms of IPNI up to one year following the surgery. Furthermore, previous studies have demonstrated that pain intensity and duration of pain influence daily activities and quality of life negatively.

Positioning of the patients on operating table is a teamwork where the operating room nurse (ORN) has a pivotal role in order to protect the patients from experiencing injuries due to e.g. nerve compression and compromised circulation. The purpose of this study is to increase the knowledge of IPNI related to positioning in patients undergoing robotic-assisted laparoscopic surgery and laparoscopic surgery. As IPNI is an unclear phenomenon that can be difficult to diagnose, we want to identify pain and other symptoms immediately after surgery that might have an impact on development of IPNI. Several studies have reported persistent pain after surgery like neuropathic pain and that neuropathic pain occur soon after nerve lesion. To get at a broader picture of IPNI we want to explore pain and other symptoms and to characterize how these symptoms might change, and to identify risk factors associated with IPNI. Therefore, the aims of the present study are:

1. Identify the incidence of IPNI up to 12 months after surgery.
2. Explore pain, other symptoms, physical function and quality of life up to 12 months after surgery.
3. Explore risk factors associated with IPNI.
4. Explore associations between IPNI and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years.
* Robotic assisted surgery and laparoscopic surgery (urological, gynecologic, gastroenterological)
* Trendelenburg with or without lithotomy positioning on operating table.
* Planned room time > 1.5 hours.
* Speak and understand Norwegian.
* Cooperate (clinical examination).

Exclusion Criteria:

* Preexisting neuropathies.
* Neurological disease.
* Impaired cognitive function.
* Drug misuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at three of the locations of Oslo University Hospital (OUS), Radium-, Ullevål- and Aker Hospital. We will include 500 patients undergoing elective robotic-assisted or laparoscopic urological, gynecologic and gastroenterological surgery in steep Trendelenburg with or without lithotomy positioning.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | 3 months
  Douleur Neuropathies (DN4) will be used to evaluate neuropathic pain. DN4 is a validated tool to screen the neuropathic origin of pain. It includes three items about the type of pain (burning/painful cold/electric shock), four items about the associated symptoms (tingling/pins and needles/numbness/itching), two about the existence of numbness in painful area (on contact/on pinching), and one about initiation or enhancement of pain rubbing. Three or more positive answers on the seven questions are defined as neuropathic pain. At baseline a study nurse will help the patients to complete the questionnaire. At follow up, for use in this study the questions are adapted for completion by the patients.
Pain | 3 months
  Brief pain inventory (BPI) will be used to measure pain occurrence, pain intensity, pain interference with function and pain relieve. Occurrence is examined using one item where the patients' ticked yes or no if they are generally bothered by pain. Three items measure pain intensity (pain now, worst pain and average pain) and seven items' measures pain interference with functioning (i.e., daily activity, mood, walking ability, normal work, sleep, enjoyment of life, relations with others). The items are scored on an 11-point numeric rating scale from 0-10. The BPI has been reported to be sensitive to change for pain intensity, and a change of two units on the 11-point scale is considered clinically significant. The BPI has been established as a reliable and valid measure of pain in a Norwegian sample.
Neuropathic symptoms | 3 months
  It is developed a study specific questionnaire about neuropathic symptoms (i.e., burning, tingling, numbness, electric shocks) as a supplement to DN4. It is also designed questions to reveal if the patients have reduced muscular force or reduced sensibility in the extremities.

SECONDARY OUTCOMES:
Physical function | 12 months
  Oswestry Disability Index (ODI) will be used to measure physical function related to pain. The ODI contains 10 items concerning intensity of pain (i.e., lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality and ability to travel). Each item is scored on a 6-point scale, with a sum score ranging from 0 (no limitation) to 100 (maximal limitation). The version 2.0 is recommended for general use, is a modification of the original ODI. ODI is a reliable and valid tool and has been translated and adapted for Norwegian patients.
Health related quality of life (Rand 12) | 12 months
  Rand 12 (SF-12 version 1) consists of 12 items; each scored on a 6-point Likert scale. The items assess eight health concepts (i.e., physical functioning, role-physical, bodily pain, general health, energy/fatigue, social functioning, role-emotional and mental health) that comprise a physical component summary (PCS) score and a mental component summary (MCS) score. It is extensively used and validated for many patient groups as well as the general population.

OTHER OUTCOMES:
Multiple symptoms (MSAS) | 12 months
  MSAS will be used to assess symptoms. The scale consist of 32 different symptoms and measure both occurrence, frequency, severity and distress. Patients indicate whether or not they had a symptom during the past week (i.e. occurrence). If yes; they are asked to rate its frequency, severity, and distress on four-to-five- point Likert scales. Scores can be utilized to aggregate subscale scores (i.e., physical and psychological) and a total score, which is the average of the 32 symptoms. The reliability and validity is well established also in Norwegian patient's samples.